CLINICAL TRIAL: NCT06531980
Title: Effektiviteten av en Digital Mestringsapp for Ungdommer Med Mild Til Moderat Angst
Brief Title: Effectiveness of a Digital Application for Adolescents With Mild to Moderate Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Bergen kommune (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 714490
Record Dates: First submitted 2024-06-28; First posted 2024-08-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Anxiety and Fear; Adolescent - Emotional Problem
Keywords: Digital Health; Digital interventions; Cognitive behavior therapy; adolescent; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: One group receives the digittal health intervention and one group receives treatment as usual
Who Masked: Investigator
Masking Description: A member of the research group will conduct the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modi-application (Experimental): 8-weeks interventions provided by the mobile application Modi. Therapist-guided intervention
  Interventions: Other: Modi
- Treatment as usual (Active Comparator): The group will receive treatment as usual.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Modi — The Modi course, an eight-week mobile application intervention for adolescents with anxiety symptoms, is based on cognitive therapy. Guided by a rule-based chatbot named "Anna," users navigate through predefined options and responses, learning about anxiety and recording their challenges. The app includes animated videos, illustrations, and audio files to enhance engagement. Modi consists of six chapters, with a focus on psychoeducation, the cognitive triangle, and exposure exercises. Participants receive guidance from two Modi therapists who provide weekly support via messages and scheduled phone calls, ensuring personalized assistance and addressing any issues throughout the course.
  Arms: Modi-application
Other: Treatment as usual — Participants receive usual treatment at their local Child and Family Services. This treatment, known as Treatment as Usual (TAU), is not standardized but reflects the care they would receive in regular practice. It aligns with national clinical guidelines and includes individual therapy, parental counseling, and assessments. Typically, the treatment is provided by a therapist trained in cognitive behavioral therapy (CBT) or a psychologist
  Arms: Treatment as usual

SUMMARY:
The goal of this randomized controlled trial is to investigate the effectiveness of a new therapist-guided rule based intervention in Bergen Municipality, Child and Family help center.

Do they have a decrease in anxiety symptoms following the intervention? Do they have an increase in functional level following the intervention?

Researchers will compare the therapist-guided rule based intervention with treatment as usual for adolescents with mild to moderate anxiety.

Participants will use the intervention, which is based on CBT, for 8 weeks.

DETAILED DESCRIPTION:
Modi is a mobile application and consists of a training program for adolescents with anxiety problems. Anxiety is one of the most common mental disorders. The anxiety symptoms usually have an age of onset in adolescence. For many, these anxiety symptoms persist into adulthood, and lead to reduced quality of life and functional impairment. The goal is to prevent anxiety disorders, comorbid disorders and loss of function as a result of the anxiety symptoms.

This study wants to investigate the effectiveness of a digital intervention in a randomized controlled trial. The study will recruit N = 128 young people aged 13-16 who will be randomized to either a therapist-guided, rule-based chatbot intervention or treatment as usual in the Child and Family Help Center in Bergen Municipality. The study will examine the clinical effects of the new intervention compared to treatment as usual

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-16
* Resides in Bergen
* Completed RCADS-25
* Reports "yes" to both questions:
* Do you have anxiety symptoms? Do you often feel stressed, scared, worried, or feel it in your body (e.g., stomach pain, heart palpitations, breathing problems, sweating, dizziness)?
* Do anxiety symptoms prevent you from doing things you want or need to do (e.g., meeting new people, giving presentations at school, going to sleepovers, going to the shopping center)? Or do you spend so much time worrying that it affects your daily life? Can read Norwegian

Exclusion Criteria:

* Currently receiving other psychological treatment
* Immediate need for other psychological treatment, such as severe depression, suicide risk, OCD, psychosis/substance abuse issues, autism spectrum disorder
* Anxiety is largely related to bullying
* Extensive school absence of more than 50% in the last three months

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Revised Child Anxiety and Depression Scale - 25 - Self-report | assessing change from screening, pre, week 2, week 4, week 6, and immediately after the intervention, follow-up 1 month, and at follow-up 6 months]
  anxiety and depressive symptoms, higher score indicates worse outcomes
Revised Child Anxiety and Depression Scale - 25 - Parent-report | assessing change from screening, pre, week 2, week 4, week 6, and immediately after the intervention, follow-up 1 month, and at follow-up 6 months]
  anxiety and depressive symptoms, higher score indicates worse outcomes

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire - Youth version | assessing change from screening, pre, week 4, immediately after the intervention, follow-up 1 month, and at follow-up 6 months]
  The scale measure adolescent's general mental health, with a higher score indicating worse symptoms. The study intends to use all three components of the measurement, including 1) the basis of SDQ, which includes 25 items on psychological attributes, 2) impact supplement, measuring functional level. The follow-up version also includes two additional follow-up questions
Strengths and Difficulties Questionnaire - Parent version | assessing change from screening, pre, week 4, immediately after the intervention, follow-up 1 month, and at follow-up 6 months]
  The scale measure parent-reported adolescent's general mental health, with a higher score indicating worse symptoms. The study intends to use all three components of the measurement, including 1) the basis of SDQ, which includes 25 items on psychological attributes, 2) impact supplement, measuring functional level. The follow-up version also includes two additional follow-up questions

OTHER OUTCOMES:
Motivation Questionnaire | week 2
  assessments of their motivation to participate in the study and interventions, developed specifically for this study
Evaluation Questionnaire | immediately after the intervention
  evaluation assessments of the Modi intervention, developed specifically for this study.
Qualitative interviews | immediately after the intervention
  Interviews with 15 adolescents from the Modi-group about their experience using the intervention
demographics | pre-intervention
  gender, age

CONTACTS AND LOCATIONS:
Overall Officials: Smiti Kahlon, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Research centre for digital mental health services, Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
The full protocol and informed consent forms are available upon request. The datasets and the statistical code will not be publicly available, but may be available upon reasonable request through correspondence with principal investigator and according to the Norwegian law and regulations.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: starting after publication
Access Criteria: PD will be made available from PI on reasonable request and according to relevant Norwegian laws and regulations